CLINICAL TRIAL: NCT07367594
Title: Comparative Evaluation of the Effect of Lavender Versus Bitter Orange Essential Oils Aromatherapy on Decreasing Dental Anxiety and Pain of Children During Administration of Local Anesthetic: (A Randomized Clinical Trial)
Brief Title: Lavender vs Bitter Orange Aromatherapy to Reduce Anxiety and Pain in Pediatric Local Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Mennatallah Khaled, general practitioner, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Menna MSA University
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Dental Anxiety; Local Anesthesia
Keywords: aromatherapy; local anesthesia injection; lavender essential oil; bitter orange essential oil; dental anxiety
MeSH Terms: interventions — lavender oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: statistician will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Lavender essential oil then Bitter Orange essential oil then Placebo (Experimental): In the first visit: Children will receive lavender essential oil in the inhaler 2 minutes before the administration of a local anesthetic agent.
  In the second visit: Children will receive bitter orange essential oil in the inhaler 2 minutes before the administration of a local anesthetic agent.
  in the third visit: Children will receive an empty inhaler 2 minutes before the administration of a local anesthetic agent.
  Interventions: Behavioral: Lavender essential oil in the inhaler; Behavioral: Bitter Orange essential oil in the inhaler; Behavioral: Epmty inhaler (Placebo)
- Arm B: Bitter Orange essential oil then Lavender essential oil then Placebo (Experimental): In the first visit: Children will receive bitter orange essential oil in the inhaler 2 minutes before the administration of a local anesthetic agent.
  In the second visit: Children will receive lavender essential oil in the inhaler 2 minutes before the administration of a local anesthetic agent.
  in the third visit: Children will receive an empty inhaler 2 minutes before the administration of a local anesthetic agent.
  Interventions: Behavioral: Lavender essential oil in the inhaler; Behavioral: Bitter Orange essential oil in the inhaler; Behavioral: Epmty inhaler (Placebo)
- Arm C: Placebo then Lavender essential oil then Bitter Orange essential oil (Active Comparator): In the first visit: Children will receive an empty inhaler 2 minutes before the administration of a local anesthetic agent.
  In the second visit: Children will receive lavender essential oil in the inhaler 2 minutes before the administration of a local anesthetic agent.
  In the third visit: Children will receive bitter orange essential oil in the inhaler 2 minutes before the administration of a local anesthetic agent.
  Interventions: Behavioral: Lavender essential oil in the inhaler; Behavioral: Bitter Orange essential oil in the inhaler; Behavioral: Epmty inhaler (Placebo)

INTERVENTIONS:
Behavioral: Lavender essential oil in the inhaler — The children will be asked to inhale the aroma (Lavender) from the inhalers for 2 minutes before local anesthetic agent injection to reduce pain and anxiety.
Behavioral: Bitter Orange essential oil in the inhaler — The children will be asked to inhale the aroma ( bitter Orange) from the inhalers for 2 minutes before local anesthetic agent injection to reduce pain and anxiety.
Behavioral: Epmty inhaler (Placebo) — The children will be asked to inhale from an empty inhaler for 2 minutes before local anesthetic agent injection.

SUMMARY:
This randomized controlled clinical trial aims to evaluate and compare the effectiveness of lavender essential oil and bitter orange essential oil aromatherapy in reducing dental anxiety and pain in children during the administration of local anesthesia. Children aged 6-12 years undergoing dental procedures requiring local anesthetic infiltration will be randomly assigned to lavender aromatherapy, bitter orange aromatherapy, or placebo (empty inhaler). Dental anxiety will be assessed using pulse rate and blood pressure measurements, while pain will be evaluated using the FLACC behavioral pain scale. The findings are expected to provide evidence on the role of aromatherapy as a non-pharmacological, safe, and cost-effective behavior guidance method in pediatric dentistry.

DETAILED DESCRIPTION:
Dental anxiety is a significant challenge in pediatric dentistry and is especially pronounced during invasive procedures such as the administration of local anesthetics. High levels of anxiety can amplify pain perception, reduce cooperation, and negatively affect the child's overall dental experience. Although pharmacological approaches such as sedation are available, they may cause undesirable side effects and are not always suitable for children. Consequently, there is increasing interest in safe, non-pharmacological alternatives such as aromatherapy, which utilizes essential plant oils to reduce anxiety and improve patient comfort.

Lavender and bitter orange essential oils have demonstrated anxiolytic and calming effects in several clinical studies, with evidence suggesting reductions in physiological stress markers such as pulse rate, blood pressure, and cortisol levels. Aromatherapy via inhalation is non-invasive, inexpensive, and well-tolerated by children. However, despite promising findings, limited research has explored and compared the clinical efficacy of different essential oils specifically in pediatric dental settings during local anesthetic injections.

This randomized controlled trial will be conducted at the Pediatric Dentistry Department, Faculty of Dentistry, MSA University. Children aged 6-12 years requiring local anesthetic infiltration will be randomly assigned to one of three groups: lavender inhalation, bitter orange inhalation, or placebo (empty inhaler). Participants will inhale the assigned aroma for 2 minutes prior to the injection. Dental anxiety will be measured using pulse oximetry and blood pressure recordings before and after the procedure, while pain will be evaluated using the FLACC scale during the injection.

The results of this study are expected to provide evidence regarding the relative effectiveness of lavender and bitter orange aromatherapy in decreasing dental anxiety and pain during anesthetic administration. The findings may support the integration of aromatherapy as a complementary, child-friendly behavior guidance technique in pediatric dental practice, promoting safer and more holistic anxiety-reduction strategies for young patients

ELIGIBILITY:
Inclusion Criteria:

* Children with the age range of 6-12 years
* Any dental procedure that requires injection of local anesthesia.
* Cooperative patients.(according to Frankl's classification class 1 and 2)
* Parents or guardians willing to participate in the study.
* Healthy child

Exclusion Criteria:

* Children with complicated systemic disease.
* Uncooperative patients. .(according to Frankl's classification class 3 and 4)
* Children with severe cognitive impairment or developmental disorders
* Children with respiratory tract infections.
* Children experiencing dental pain such as (acute pain or hyperemia).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety level (objective) | baseline (5 minutes before session), during injection (real time), and immediately post injection (within 5 minutes)
  tool: pulse oximeter unit: beats per minute

SECONDARY OUTCOMES:
anxiety level (objective) | immediately before the injection (baseline), immediately after the injection (post injection)
  tool: digital blood pressure monitor, unit: systolic/diastolic mmhg
pain assessment | during the injection
  assessment of pain by FLACC (face-leg-activity-cry-consolability) scale score (0-2) (0 is the best outcome) (2 is the worst)

CONTACTS AND LOCATIONS:
Locations (1):
- October University for Modern Science and Art, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes